CLINICAL TRIAL: NCT01616472
Title: WEUKBRE5716: Quantifying the Burden of Steroid-related Damage in Systemic Lupus Erythematosus in the Hopkins Lupus Cohort
Brief Title: WEUKBRE5716: Steroid-related Damage in Systemic Lupus Erythematosus (Hopkins)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116015; WEUKBRE5716 (Other: GSK)
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: hypertension; avascular necrosis; systemic lupus erythematosus; osteoporosis; Steroid; diabetes; cataracts
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Hypertension; Osteonecrosis; Osteoporosis; Diabetes Mellitus; Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- Incident diabetes cases: Individuals with newly diagnosed SLE selected from the Hopkins Lupus Cohort (1987-2011) who are newly diagnosed with diabetes during follow-up, subsequent to SLE diagnosis.
  Interventions: Drug: Cumulative corticosteroid exposure
- Incident diabetes controls: Individuals with newly diagnosed SLE selected from the Hopkins Lupus Cohort (1987-2011) who have no record of diabetes during follow-up time (years) since SLE diagnosis that is equivalent to length of case at-risk time. Controls are matched to cases on decade of SLE diagnosis: 1987-1989, 1990-1999, 2000-2009, 2010+
  Interventions: Drug: Cumulative corticosteroid exposure
- Incident hypertension cases: Individuals with newly diagnosed SLE selected from the Hopkins Lupus Cohort (1987-2011) who are newly diagnosed with hypertension during follow-up, subsequent to SLE diagnosis.
  Interventions: Drug: Cumulative corticosteroid exposure
- Incident hypertension controls: Individuals with newly diagnosed SLE selected from the Hopkins Lupus Cohort (1987-2011) who have no record of hypertension during follow-up time (years) since SLE diagnosis that is equivalent to length of case at-risk time. Controls are matched to cases on decade of SLE diagnosis: 1987-1989, 1990-1999, 2000-2009, 2010+
  Interventions: Drug: Cumulative corticosteroid exposure
- Incident cataract cases: Individuals with newly diagnosed SLE selected from the Hopkins Lupus Cohort (1987-2011) who are newly diagnosed with cataract during follow-up, subsequent to SLE diagnosis.
  Interventions: Drug: Cumulative corticosteroid exposure
- Incident cataract controls: Individuals with newly diagnosed SLE selected from the Hopkins Lupus Cohort (1987-2011) who have no record of cataract during follow-up time (years) since SLE diagnosis that is equivalent to length of case at-risk time. Controls are matched to cases on decade of SLE diagnosis: 1987-1989, 1990-1999, 2000-2009, 2010+
  Interventions: Drug: Cumulative corticosteroid exposure
- Incident osteoporosis cases: Individuals with newly diagnosed SLE selected from the Hopkins Lupus Cohort (1987-2011) who are newly diagnosed with osteoporosis during follow-up, subsequent to SLE diagnosis.
  Interventions: Drug: Cumulative corticosteroid exposure
- Incident osteoporosis controls: Individuals with newly diagnosed SLE selected from the Hopkins Lupus Cohort (1987-2011) who have no record of osteoporosis during follow-up time (years) since SLE diagnosis that is equivalent to length of case at-risk time. Controls are matched to cases on decade of SLE diagnosis: 1987-1989, 1990-1999, 2000-2009, 2010+
  Interventions: Drug: Cumulative corticosteroid exposure
- Incident avascular necrosis cases: Individuals with newly diagnosed SLE selected from the Hopkins Lupus Cohort (1987-2011) who are newly diagnosed with avascular necrosis during follow-up, subsequent to SLE diagnosis
  Interventions: Drug: Cumulative corticosteroid exposure
- Incident avascular necrosis controls: Individuals with newly diagnosed SLE selected from the Hopkins Lupus Cohort (1987-2011) who have no record of avascular necrosis during follow-up time (years) since SLE diagnosis that is equivalent to length of case at-risk time. Controls are matched to cases on decade of SLE diagnosis: 1987-1989, 1990-1999, 2000-2009, 2010+
  Interventions: Drug: Cumulative corticosteroid exposure

INTERVENTIONS:
Drug: Cumulative corticosteroid exposure — Cumulative steroid exposure will be modeled as cumulative dose (prednisone equivalent mg), cumulative days of exposure at any dose, cumulative days of exposure to doses ≥7.5mg and cumulative days of exposure to doses ≥20mg.

SUMMARY:
The study is designed to assess the association between steroid exposure and five potentially steroid-related adverse events within a cohort of individuals with systemic lupus erythematosus (SLE). Study objectives are to quantify the fraction of the risk of new (i) diabetes, (ii) hypertension, (iii) cataracts, (iv) osteoporosis and (v) avascular necrosis that is attributable to cumulative corticosteroid exposure in SLE patients. The study will consist of five matched case-control analyses nested within the Hopkins Lupus Cohort. Cases will be incident SLE cases who have developed one of the case outcomes (diabetes, hypertension, cataracts, osteoporosis with fracture or vertebral collapse or avascular necrosis). Controls will be matched to cases on time since SLE diagnosis. The primary exposures to be assessed are cumulative dose of steroid (g) and cumulative duration of exposure to steroids. The extent of the risk associated with steroids will be explored through modeling of the relationship and through calculation of attributable risks of exposure (number of cases associated with the highest exposure quartile of each primary exposure).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed SLE as per ACR criteria
* No history of "case" event of interest in follow-up time prior to SLE diagnosis (case) or during follow-up time since SLE diagnosis that is equivalent to length of case at-risk time period (controls)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases and controls will be identified from the Hopkins Lupus Cohort, a prospective longitudinal study of lupus activity, organ damage, and quality of life in patients with SLE which has followed patients up since 1987. The cohort database is continually updated and includes socio-demographic information, medical and reproductive history, comorbidities, SLE complications, and treatment. Data, collected at each patient visit, includes SLE clinical activity indices, laboratory data and treatment (medication and dose).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
New diagnoses of diabetes, hypertension, cataracts, osteoporosis, or avascular necrosis | Over a period of 25 years from 1987-2011
  New diagnoses of diabetes, hypertension, cataracts, osteoporosis, or avascular necrosis recorded after SLE diagnosis in the Hopkins Lupus cohort

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Davidson JE, Fu Q, Rao S, Magder LS, Petri M. Quantifying the burden of steroid-related damage in SLE in the Hopkins Lupus Cohort. Lupus Sci Med. 2018 May 14;5(1):e000237. doi: 10.1136/lupus-2017-000237. eCollection 2018. PMID 29765616